CLINICAL TRIAL: NCT01180673
Title: Counseling Older Adults to Control Hypertension
Acronym: COACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-416; P60MD000206 (NIH)
Record Dates: First submitted 2010-07-27; First posted 2010-08-12 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Hypertension; Older Adults; Motivational Interviewing; Lifestyle Counseling; Senior Centers
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINT-TLC (Experimental)
  Interventions: Behavioral: MINT-TLC
- Control Condition (Active Comparator)
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: MINT-TLC — This intervention is based on established clinical practice guidelines for prevention and treatment of hypertension, which recommend weight loss (if overweight), limiting sodium and alcohol intake, regular physical activity, and eating a low-fat diet that is rich in fruit and vegetables. Seniors will attend weekly group classes conducted by trained research assistants for the first 12 weeks (intensive phase); followed by three individual motivational interview (MINT) sessions that will occur monthly over the next three months (extended phase); and finally each senior will receive three bi-monthly booster MINT sessions in the remaining six months (maintenance phase).
  Arms: MINT-TLC
Behavioral: Control Condition — Seniors randomized to the control arm will receive a single individual brief advice session on therapeutic lifestyle changes recommended for blood pressure reduction. In addition, they will be given print versions of the NHLBI publications "Your Guide to Lowering Blood Pressure"; and "Facts about the DASH Eating Plan." Sessions will be delivered by trained research assistants.
  Arms: Control Condition

SUMMARY:
This study will evaluate the effect of a senior center-based comprehensive therapeutic lifestyle intervention delivered through group-based counseling and motivational interviewing (MINT-TLC) among 250 hypertensive African American or Latino seniors age 60 and older in a randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Diagnosis of HTN
* Taking at least one anti-hypertensive medication
* Self-identified Black, African American, or Latino

Exclusion Criteria:

* Unable to comply with the study protocol
* Participation in other hypertension studies
* Severe hearing impairment
* Severe visual impairment
* Arm circumference > 42 cm for large cuff, or arm circumference > 52 cm for extra large cuff (if extra large cuff is available)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Within-individual change in systolic blood pressure and diastolic blood pressure from baseline to 12 months | 12 months

SECONDARY OUTCOMES:
Change in physical activity level from baseline to 12 months | 12 months
  Physical activity is assessed using the Yale Physical Activity Scale (YPAS) and the International Physical Activity Questionnaire (IPAQ). Data collected with the YPAS will be reported as a final total activity dimension score. Data collected for the IPAQ will be expressed in MET-min per day or categorically (low, moderate, high).
Percent change in weight from baseline to 12 months | 12 months
Change in number of daily servings of fruits and vegetables from baseline to 12 months | 12 months
Proportion of participants with adequate blood pressure control at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olugbenga Ogedegbe, MD, MS, MPH, FACP, Principal Investigator — NYU Langone Health
Locations (1):
- Senior Centers affiliated with NYC Department for the Aging, New York, New York, United States

REFERENCES:
- [Derived] Ogedegbe G, Fernandez S, Fournier L, Silver SA, Kong J, Gallagher S, de la Calle F, Plumhoff J, Sethi S, Choudhury E, Teresi JA. The Counseling Older Adults to Control Hypertension (COACH) trial: design and methodology of a group-based lifestyle intervention for hypertensive minority older adults. Contemp Clin Trials. 2013 May;35(1):70-9. doi: 10.1016/j.cct.2013.02.008. Epub 2013 Feb 24. PMID 23462343